CLINICAL TRIAL: NCT00914030
Title: Visual Exploration and Attention : Studies in Patients With Schizophrenia and Autism Spectrum Disorders
Brief Title: Visual Exploration and Attention: Studies in Patients With Schizophrenia and Autism Spectrum Disorders
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2008-A01459-46
Record Dates: First submitted 2009-06-02; First posted 2009-06-04 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Autism Spectrum Disorders; Schizophrenia
Keywords: Visual perception; Local/global processing; Attention; Visual priming; Collinearity; Grouping
MeSH Terms: conditions — Autism Spectrum Disorder; Schizophrenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- A1: Patients with schizophrenia
  Interventions: Other: Neuropsychological evaluation
- A2: Control subjects matched individually with patients with schizophrenia
  Interventions: Other: Neuropsychological evaluation
- B1: Adult subjects with autism
  Interventions: Other: Neuropsychological evaluation
- B2: Control subjects matched individually with adult subjects with autism
  Interventions: Other: Neuropsychological evaluation
- C1: Children with autism
  Interventions: Other: Neuropsychological evaluation
- C2: Control subjects matched individually with children with autism
  Interventions: Other: Neuropsychological evaluation

INTERVENTIONS:
Other: Neuropsychological evaluation — Study one: global/local processing, with a neutral prime (stimulus influencing the processing of the subsequent stimulus)Study two: global/ local processing with a prime whose elements are collinear.Study three: global/local processing with a prime whose elements are not collinear
  Other Names: Each study will be conducted successively in each group (A1/ A2, B1/B2, C1/C2).

SUMMARY:
The aim of the protocol is to better understand the impairments in visual processing, as such impairments may induce social interaction difficulties in subjects with autism spectrum disorders (adults and children) and schizophrenia, like face exploration.The same protocol will be used for the three populations, each population being compared with matched controls. The explorations are designed to test two different hypotheses regarding the mechanisms of the visual perception difficulties of the two populations. Even though difficulties to extract the global form of objects have been described in both subjects with autism and schizophrenia, we will test two different hypotheses for the two populations. We will test the hypothesis that subjects with autism display an advantage for the processing of local information arising at an early level of processing, whereas disorders observed in patients with schizophrenia originate from attention disorders. The protocol includes three consecutive studies, each one being applied in each of the three populations.

ELIGIBILITY:
Inclusion Criteria:

* IQ above 70, as evaluated with the WAIS III in adults and with the WISC in children
* signed consent
* DSM IV criteria in case of autism spectrum disorders or schizophrenia

Exclusion Criteria:

* grave or non stabilized somatic pathology
* pathology affecting the central nervous system; other than the studied pathologies
* intake of psychotropic drug, except for patients
* invalidating sensory processes

Ages: 7 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Psychiatry clinic in Strasbourg and Brumath. Pedopsychiatry Clinic in Strasbourg. Residents of Strasbourg and Brumath
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2009-06; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Anne GIERSCH, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (5):
- France (5):
  - Pôle départemental du Centre de Ressources Autisme pour adultes (67) - Etablissement public de santé Alsace-Nord (site de Brumath), Brumath
  - Centre de Ressources Autisme Pôle adultes (68) - Espace Autisme 68, Colmar
  - Clinique Lautréamont, Loos
  - Pôle régional du Centre de Ressources Autisme pour enfants et adolescents - Unité d'évaluation des troubles du développement Hôpital de l'Elsau - Pôle de Psychiatrie - Unité d'évaluation des troubles du développement Hôpital de l'Elsau - HUS, Strasbourg
  - INSERM U666 ; Pôle de Psychiatrie - Service de Psychiatrie Adulte- HUS, Strasbourg